CLINICAL TRIAL: NCT04052594
Title: A Randomized, Double-Blind, Single Dose, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3475766
Brief Title: A Study of LY3475766 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17394; J1T-MC-GZEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04-15

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3475766 - IV (Experimental): LY3475766 administered intravenously (IV) to participants with dyslipidemia
  Interventions: Drug: LY3475766 - IV
- Placebo - IV (Placebo Comparator): Placebo administered IV to participants with dyslipidemia
  Interventions: Drug: Placebo - IV
- LY3475766 - SC (Experimental): LY3475766 administered subcutaneously (SC) to participants with dyslipidemia
  Interventions: Drug: LY3475766 - SC
- Placebo - SC (Placebo Comparator): Placebo administered SC to participants with dyslipidemia
  Interventions: Drug: Placebo - SC

INTERVENTIONS:
Drug: LY3475766 - IV — Administered IV
  Arms: LY3475766 - IV
Drug: LY3475766 - SC — Administered SC
  Arms: LY3475766 - SC
Drug: Placebo - IV — Administered IV
  Arms: Placebo - IV
Drug: Placebo - SC — Administered SC
  Arms: Placebo - SC

SUMMARY:
This study will evaluate the safety and tolerability of LY3475766 when given to participants with high levels of blood fat called triglycerides. It will also investigate how the body processes the study drug and the effect of the study drug on the body. Information about any side effects will be documented. This study will last up to 16 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, apart from dyslipidemia
* Male participants must agree to adhere to contraception restrictions
* Female participants must be of nonchildbearing potential and include those who are infertile due to surgical sterilization or those who are postmenopausal
* Have a body mass index (BMI) >18.5 and <40 kilograms per meter squared (kg/m²)
* Have clinical laboratory test results within normal reference range, or acceptable deviations per investigator discretion
* Have a fasting triglyceride (TG) level that is 135 to 499 milligrams per deciliter (mg/dL), inclusive, at both screening and Day -1
* Have a fasting low density lipoprotein cholesterol (LDL-C) level greater than or equal to (≥) 70 mg/dL, inclusive, at screening and Day -1
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight change)
* Have not modified diet or adopted any nutritional lifestyle modification within 3 months prior to randomization

Exclusion Criteria:

* Are taking or have started taking Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors within 3 months prior to randomization; or statins, fibrates, or niacin ≤1000 mg/day within 8 weeks prior to randomization; or niacin >1000 milligrams per day (mg/day) within 16 weeks prior to randomization; or any other lipid-lowering agents within 1 month prior to randomization
* Are taking or have started taking a beta-blocker, antiarrhythmic, non-dihydropyridine calcium channel blocker, ivabradine, or any other heart rate lowering agent within 1 month or 5 half-lives prior to randomization, whichever is longer
* Have a diagnosis of diabetes mellitus (type 1 diabetes mellitus or type 2 diabetes mellitus) or have 1 of the following at screening: fasting plasma glucose concentration ≥126 mg/dL (7.0 millimoles per liter [mmol/L]) OR a glycated hemoglobin level ≥6.5% (48 millimoles per mole [mmol/mol])
* Have previously completed or withdrawn from this study or any other study investigating LY3475766, and have previously received the investigational product
* Have known allergies to LY3475766, related compounds, or any components of the formulation, or history of significant atopy
* Have a seated heart rate ≤50 beats per minute
* Have clinically significant abnormal electrocardiogram (ECG) results constituting a risk while taking the investigational product, as determined by the investigator
* Have an abnormal blood pressure (BP) as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 85
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3475766 | Predose up to Day 85
  PK: AUC of LY3475766
PK: Maximum Observed Drug Concentration (Cmax) of LY3475766 | Predose up to Day 85
  PK: Cmax of LY3475766
PK: Time to Maximum Observed Drug Concentration (Tmax) of LY3475766 | Predose up to Day 85
  PK: Tmax of LY3475766
Pharmacodynamics (PD): Percent Change from Baseline in Triglycerides (TG) | Baseline, Day 85
  PD: Percent Change from Baseline in TG
PD: Percent Change from Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline, Day 85
  PD: Percent Change from Baseline in LDL-C
PD: Percent Change from Baseline in Apolipoprotein B (ApoB) | Baseline, Day 85
  PD: Percent Change from Baseline in ApoB

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - WCCT Global, Cypress, California
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance Dallas, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaudet D, Gonciarz M, Shen X, Leohr JK, Beyer TP, Day JW, Mullins GR, Zhen EY, Hartley M, Larouche M, Konrad RJ, Benichou O, Ruotolo G. Targeting the angiopoietin-like protein 3/8 complex with a monoclonal antibody in patients with mixed hyperlipidemia: a phase 1 trial. Nat Med. 2025 Aug;31(8):2632-2639. doi: 10.1038/s41591-025-03830-4. Epub 2025 Jul 10. PMID 40640392